CLINICAL TRIAL: NCT01971268
Title: Marginal Bone Behavior of Dental Implants to Different Rehabilitation Protocols
Brief Title: Compare the Success Rate of T3 Dental Implant (Biomet 3I) With or Without Platform-switch Concept
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Implantology Institute (Other)
Responsible Party: Principal Investigator, Andre Chen, Mcs, Implantology Institute
Other Study IDs: II-02
Record Dates: First submitted 2013-10-17; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Implants; Bone Loss
Keywords: T3 dental implants; Marginal bone loss; Survival rate
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Platform-Switch Group: T3 dental implant, with platform-switch dental implant platform concept, measure marginal bone loss
  Interventions: Device: Dental Implant; Device: Platform-Switch Dental Implant
- Platform-Matched Group: T3 dental implant, platform-matched dental implant platform concept, measure marginal bone loss
  Interventions: Device: Dental Implant; Device: Platform-Matched dental implant

INTERVENTIONS:
Device: Dental Implant — place dental implants according to manufacturer guidelines
  Other Names: Biomet 3i T3 dental implant
Device: Platform-Switch Dental Implant — Place Dental Implant with an abutment narrower than the implant platform
  Other Names: Biomet 3I Dental Implant Platform-Switch; Discrepant Platform implant; non-matched dental implant
  Groups: Platform-Switch Group
Device: Platform-Matched dental implant — Place Dental Implant with abutment with same size as the platform
  Other Names: Biomet 3I T3 Dental Implant; non-discrepant platform dental implant
  Groups: Platform-Matched Group

SUMMARY:
In patients that received a T3 (Biomet 3I) dental implant, does the use of platform-switch concept compared to the use of platform-matched concept, refrain marginal bone loss during osseointegration phase (t=12 weeks =T1) and from then to final rehabilitation (t= placement of the final restoration = at 18 weeks=T2)

DETAILED DESCRIPTION:
Patients from a private practice who received dental implants (T3 dental implant Biomet 3I) from November 2012 to October 2013 were eligible to enter the study.

Two groups were formed: one group received a T3 dental implant with platform switch concept and the other received an implant with platform matched type of connection.

We evaluate osseointegration at T1 (12 weeks) and marginal bone position in relation to the implant platform at baseline (implant installation) T0 and again at T1 and T2.

From data recorder in T0,T1 and T2, we evaluate changes in marginal bone position.

ELIGIBILITY:
Inclusion Criteria:

* Single unit implant rehabilitation
* Maxilla and mandible
* Biomet 3I T3 dental implant placed
* Final Rehabilitation placed

Exclusion Criteria:

* Immediate implants
* Radiographic impossibility of measure
* Absence of baseline T0 radiograph
* Smoking habits (more 10 cigarets a day)
* Diabetes
* Patients who receive Radio or/and Chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population from a private office who seek care to replace missing teeth, must have economical status to do implant supported rehabilitations
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-08 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Position of Implant Platform to marginal bone | At Baseline (T0)
  Compare marginal bone position at baseline T0 (measured radiographically (digital) from the most coronal position of marginal bone to the most coronal position of the platform, measured in the most mesial and distal part (two measures) of the implant platform.
Marginal Bone Position at 8 Weeks | At 12 weeks (T1) after Baseline
  Compare marginal bone position at T1, 12 weeks after baseline (T0) (measured radiographically (digital) from the most coronal position of marginal bone to the most coronal position of the platform, measured in the most mesial and distal part (two measures) of the implant platform
Marginal Bone Position at 12 Weeks | At 18 Weeks (T2) after baseline (T0)
  Compare marginal bone position at T2, 18 weeks from baseline (T0) (measured radiographically (digital) from the most coronal position of marginal bone to the most coronal position of the platform, measured in the most mesial and distal part (two measures) of the implant platform.

SECONDARY OUTCOMES:
Osseointegration | At 12 weeks
  measure the ability of the implant to integrate in bone

CONTACTS AND LOCATIONS:
Overall Officials: Andre Chen, Msc, Principal Investigator — Implantology Institute; João Caramês, Phd, Study Director — Implantology Institute; Helena Francisco, Msc, Study Chair — Implantology Institute; Elena Cervino, Msc, Study Chair — Implantology Institute
Locations (1):
- Instituto de Implantologia, Lisbon, Lisbon District, Portugal